CLINICAL TRIAL: NCT06536439
Title: Planning Operative Strategy Using a Digital Renal Artery Clamping Tool: a Randomized Controlled Trial Evaluating the DIPLANN 3D Model for Selective Arterial Clamping During Robot-Assisted Partial Nephrectomy
Brief Title: Planning Operative Strategy Using a Digital Renal Artery Clamping Tool
Acronym: PODRACING
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Stichting tegen Kanker (Other); University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONZ-2023-0558
Record Dates: First submitted 2024-07-15; First posted 2024-08-05 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Kidney Cancer; Kidney Neoplasms; Kidney Diseases; Renal Cancer; Renal Cell Carcinoma; Renal Disease
Keywords: Kidney Cancer; Renal Cell Carcinoma; Minimally Invasive Surgery; Robot-Assisted Surgery; Robot-Assisted Partial Nephrectomy; RAPN; 3D; Perfusion Zone
MeSH Terms: conditions — Kidney Neoplasms; Kidney Diseases; Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: Confirmatory, multicentric, unblinded, randomized, controlled, pivotal trial using parallel group assignment and stratified randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- DIPLANN-tool + conventional CT imaging (Experimental): Pre-operative planning and peri-operative guidance with DIPLANN-tool and conventional CT imaging.
  Interventions: Device: Pre-operative explanation of the procedure (DIPLANN + CT); Device: Pre-operative surgical planning (DIPLANN + CT); Procedure: RAPN (DIPLANN + CT)
- Conventional CT imaging alone (Active Comparator): Pre-operative planning and peri-operative guidance with conventional CT imaging alone (standard of care).
  Interventions: Device: Pre-operative explanation of the procedure (CT only); Device: Pre-operative surgical planning (CT only); Procedure: RAPN (CT only)

INTERVENTIONS:
Device: Pre-operative explanation of the procedure (DIPLANN + CT) — Pre-operative study visit explaining the RAPN procedure using the 3D model / DIPLANN-tool (with or without classical CT imaging). Included in this visit is a pre-operative physical examination (height, weight, abdominal examination), pre-operative blood examination (Hb, creatinin, eGFR) and patient questionnaires regarding patient knowledge, patient anxiety and patient quality of life.
  Arms: DIPLANN-tool + conventional CT imaging
Device: Pre-operative surgical planning (DIPLANN + CT) — Online assessment by surgeon regarding clamping strategy. Assisted by DIPLANN-tool + CT scan.
  Arms: DIPLANN-tool + conventional CT imaging
Procedure: RAPN (DIPLANN + CT) — Robot-assisted partial nephrectomy surgical procedure. Peri-operative guidance by DIPLANN-tool + CT scan.
  Arms: DIPLANN-tool + conventional CT imaging
Device: Pre-operative explanation of the procedure (CT only) — Pre-operative study visit explaining the RAPN procedure using CT imaging alone. Included in this visit is a pre-operative physical examination (height, weight, abdominal examination), pre-operative blood examination (Hb, creatinin, eGFR) and patient questionnaires regarding patient knowledge, patient anxiety and patient quality of life.
  Arms: Conventional CT imaging alone
Device: Pre-operative surgical planning (CT only) — Online assessment by surgeon regarding clamping strategy. Assisted by classical CT imaging only.
  Arms: Conventional CT imaging alone
Procedure: RAPN (CT only) — Robot-assisted partial nephrectomy surgical procedure. Peri-operative guidance by CT imaging only.
  Arms: Conventional CT imaging alone

SUMMARY:
A proposed new tool ('DIPLANN-tool' - Digital Planning in Nephrectomy) for predicting kidney perfusion zones on a segmented 3D model during robot-assisted partial nephrectomy (RAPN) for localized renal cancer demonstrated high accuracy when planning selective clamping (SC) for RAPN. However, the tool's clinical added value still needs to be confirmed. Therefore, a randomized controlled trial using a study and control group is the preferred study design.

Experimental group: the use of the DIPLANN-tool + conventional computed tomography (CT) imaging for preoperative planning and perioperative guidance during RAPN.

Control group: the use of only conventional CT imaging for preoperative planning and perioperative guidance during RAPN (= current standard of care).

The primary endpoint is planning and performing as planned a SC strategy. Secondary endpoints include patients' health, patients' insight and surgeons' benefits.

DETAILED DESCRIPTION:
BACKGROUND:

For patients diagnosed with localized kidney cancer, two main options exist to surgically remove the kidney tumor. During radical nephrectomy (RN), the entire kidney is removed. During partial nephrectomy (PN), only the tumor is resected, safeguarding the function of the remaining healthy kidney tissue. This last procedure is preferred, but not always technically feasible. To resect only the tumor, a balance has to be found in the clamping approach: clamping the blood supply to the kidney assures bloodless tumor resection, yet compromises the postoperative renal function due to the temporary ischemia. Tumor resection without clamping on the other hand, might lead to substantial blood loss. That is why "selective clamping" (SC) is proposed. In this approach, only those selective arteries are clamped that perfuse the zone including the tumor. The main drawback of this strategy is that it is often not clear which arteries should be clamped based on standard preoperative imaging, while misjudgment can lead to a high-risk surgery with excessive bleeding or prolonged ischemia time. Therefore, RN is currently recommended when PN is considered not feasible. Better prediction of individual kidney perfusion will allow to perform more frequently a PN and thus save healthier kidney tissue. Additionally, it is difficult for patients to assess their own individual oncological situation based on 2D CT images.

With this project, the investigators want to offer the surgeon an easy-to-use virtual planning tool that facilitates the decision-making process regarding the feasibility of PN and the corresponding optimal clamping strategy. This tool uses virtual 3D models based on CT scans, to visualize precise information on the different anatomical structures and perfusion zones. This may also improve patients' understanding of their own individual situation. The proposed new tool (DIPLANN-tool) for predicting kidney perfusion zones on a segmented 3D model during robot-assisted partial nephrectomy (RAPN) for localized renal cancer demonstrated high accuracy when planning selective clamping (SC) for RAPN. However, the tool's clinical added value still needs to be confirmed. Therefore, a randomized controlled trial using a study and control group is the preferred study design.

DESIGN:

A confirmatory, multicentric, unblinded, randomized, controlled, pivotal trial using parallel group assignment and stratified randomization.

Experimental group: the use of the DIPLANN model + conventional CT imaging for preoperative planning and perioperative guidance.

Control group: the use of only conventional CT imaging for preoperative planning and perioperative guidance (= current standard of care).

METHODOLOGY:

Sample size calculation: 235 patients.

Patients will be randomized according to a 1:1 allocation ratio to either the experimental group (the DIPLANN-tool in combination with conventional CT imaging) or the control group (conventional CT imaging alone), using permuted block randomization with blocks of varying size.

Randomization will be stratified on the following variables:

* Whether SC is deemed possible according to the DIPLANN-tool in combination with conventional CT imaging or on conventional CT imaging alone, as assessed by an independent surgeon (between inclusion and randomization) who will not be not involved in the RAPN surgical procedure (yes vs no).
* Hospital where surgery is performed.
* PADUA classification (low (<8) and intermediate (8-9) vs high-risk (>9)). In case of multiple masses, the mass with the highest individual PADUA classification will be used.

PRIMARY OBJECTIVE:

To assess if the DIPLANN-tool in combination with conventional CT imaging is superior to conventional CT imaging alone, with respect to planning and performing as planned a SC strategy during RAPN, in patients diagnosed with localized kidney cancer who are planned to undergo renal cancer surgery and in whom SC is deemed possible either according to the DIPLANN-tool in combination with conventional CT imaging or according to conventional CT imaging only, as assessed between inclusion and randomization by an independent surgeon.

SECONDARY OBJECTIVES:

* To assess if the DIPLANN-tool in combination with conventional CT imaging is superior to conventional CT imaging alone, with respect to planning and performing as planned a SC strategy during RAPN, in patients diagnosed with localized kidney cancer who are planned to undergo renal cancer surgery.
* To compare the DIPLANN-tool in combination with conventional CT imaging to conventional CT imaging alone with respect to: patients' health, patients' insight, and surgeons' benefits.

ENDPOINTS:

The primary endpoint is planning and performing as planned a SC strategy. Secondary endpoints include patients' health, patients' insight and surgeons' benefits.

Extended listing of all outcome measures: see below.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or above
* cT1-2 N0 M0 renal mass
* planned to undergo RAPN
* multiphase CT scan with arterial phase available
* voluntary given and written informed consent
* sufficient in at least one of the study languages: Dutch, English, French

For the primary objective, SC needs to be deemed possible either according to the DIPLANN-tool in combination with conventional CT imaging or according to conventional CT imaging only, as assessed by an independent surgeon (between inclusion and randomization) who will not be involved in the RAPN surgical procedure, in order to be included in the analysis set. On the DIPLANN tool, SC is deemed feasible if >= 90% tumor ischemia and <= 70% renal parenchyma ischemia can be achieved. If these criteria are met, but it is technically or anatomically not feasible according to the independent surgeon to perform SC, he can deviate from these criteria and thus claim SC is not deemed possible. The results for the total population (patients in which SC is deemed possible AND impossible pre-operatively by an independent surgeon) will also be analyzed as a secondary objective.

Exclusion Criteria:

* > 3 ipsilateral renal masses
* women who are pregnant or breastfeeding
* previous renal surgery that is expected to complicate renal cancer surgery
* cT ≥ 3
* planned off-clamp resection
* cognitive disorder which impedes with completing study questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 235 (Estimated)
Dates: Start 2024-06-27 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Selective clamping | During surgery
  Planning and performing as planned a selective clamping (SC) strategy (considered by the surgeon at the end of surgery, objectified pre- and postoperatively through online assessment on study website and controlled through video-analysis): planning SC and performing the planned SC strategy = positive outcome; planning SC and performing another SC strategy or full clamping (FC) = negative outcome; planning FC = negative outcome.

SECONDARY OUTCOMES:
eGFR 6 months | 6 months postoperatively
  Change in eGFR at 6 months after surgery compared to eGFR preoperatively.
Clamping strategy | During surgery
  Clamping strategy performed (selective clamping or full clamping).
Hilar dissection time | During surgery
  Time to dissect hilum (minutes) as analyzed on postoperative surgical video analysis.
Conversion to full clamp | During surgery
  Conversion from SC to FC.

OTHER OUTCOMES:
Complications | 90 days postoperatively
  Intra-operative and 90-day postoperative complications.
Estimated blood loss | During surgery
  Estimated blood loss during surgery (mL).
Perfusion model validation | During surgery
  Concordance between 3D perfusion model and peroperative kidney surface perfusion as visualized by ICG as estimated by postoperative surgical video analysis.
Low eGFR 6 months | 6 months postoperatively
  eGFR (CKD-EPI) <45 ml/min at 6 months after surgery.
Postoperative eGFR | up to 12 months postoperatively
  Change in eGFR (CKD-EPI) after surgery at other time points up to 1 year (postoperative day 1, last measurement before discharge, postoperatively 1 month, 3 months, 12 months) compared to eGFR preoperatively.
Ischemia time | During surgery
  Ischemia time during surgery (seconds).
Positive surgical margin rate | Postoperatively on average 10 days after surgery
  Positive surgical margin (PSM), as analyzed on histopathological examination.
Console time | During surgery
  Robotic console time of surgery (minutes).
Hospital stay | From day of surgery to day of discharge from the hospital: number of days includes day of the surgery as the first day and day of discharge from the hospital as the final day (estimated at 3 days, longer if more complicated hospitalisation)
  Length of hospital stay after surgery (days).
Patient quality of life | up to 12 months postoperatively
  Quality of life (according to the European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire: higher score = worse quality of life) up until 1 year after surgery (preoperatively, postoperatively at 3 months, 6 months, 12 months).
Anxiety 1 | Preoperatively
  Preoperative anxiety for surgery questionnaire: Hospital Anxiety and Depression Scale (HADS): higher score = more anxiety.
Anxiety 2 | Preoperatively
  Preoperative anxiety for surgery questionnaire: Symptom Distress Thermometer (SDT): higher score = more anxiety.
Patient knowledge | Preoperatively
  Preoperative patient knowledge questionnaire. Higher score = more knowledge.
Kidney dissection time | During surgery
  Time to dissect kidney (minutes) as analyzed on postoperative surgical video analysis.
Superselective clamping rate | During surgery
  Superselective clamping (yes/no) as analyzed on postoperative surgical video analysis.
Ischemic renal parenchyma | During surgery
  Percent renal parenchyma rendered ischemic.
Conversion rate | During surgery
  Conversion from partial to radical nephrectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Van Praet, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (5):
- Belgium (5):
  - AZORG, Aalst
  - AZ Sint-Jan, Bruges
  - ZOL, Genk
  - AZ Maria Middelares, Ghent
  - Ghent University Hospital, Ghent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vangeneugden J, Vermijs S, De Backer P, Hemeryck B, Berquin C, De Visschere P, Decaestecker K, Debbaut C, Van Praet C. Three-dimensional Perfusion-zone Models Allow More Selective Clamping During Robot-assisted Partial Nephrectomy: Brief Report on a Retrospective Analysis. Eur Urol Open Sci. 2025 Nov 5;82:128-130. doi: 10.1016/j.euros.2025.10.013. eCollection 2025 Dec. PMID 41280160